CLINICAL TRIAL: NCT06110780
Title: Investigation of the Hemodynamic, Cardioprotective and Anti-inflammatory Effectiveness of Electroacupuncture in Patients Undergoing Coronary Artery Bypass Surgery: Randomized, Controlled Study.
Brief Title: Investigation of the Effectiveness of Electroacupuncture in Patients Undergoing Coronary Artery Bypass Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Associate professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022/01
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Protective Effects of Acupuncture in Cardiac Surgery
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture group (Active Comparator): The conductor of the study, an acupuncturist experienced in electroacupuncture, will apply electroacupuncture to the PC 6, LU7, LU2 points for 30 minutes on the day before surgery and on the day of surgery.
  The placement of the needles will be applied to a depth of 1-2 cm, depending on the thickness of the local tissues, according to Traditional Chinese Medicine standards.
  The EA parameter will be set to a frequency of 2 HZ/100 HZ at a current that the patients' tolerance is best within the range of 0.5 mA to 1.2 mA.
  The patient will be electrically stimulated for 30 minutes until the patient feels "Teh Chi" - "heaviness, numbness and swelling".
  Interventions: Other: acupuncture
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: acupuncture — The insertion of the needles will be applied to a depth of 1-2 cm according to the thickness of the local tissues according to the standards of Traditional Chinese Medicine. The EA parameter will be set to a frequency of 2 HZ/100 HZ at a current that the patients' tolerance is best between 0.5 mA and 1.2 mA.
  The patient will be electrically stimulated for 30 minutes until the patient feels "Teh Chi" - "heaviness, numbness and swelling".
  Arms: Acupuncture group

SUMMARY:
In China, acupuncture has been used for nearly 5,000 years to treat diseases and symptoms.

Increasing evidence suggests that acupuncture, acupressure, and electroacupuncture (EA) may be useful in treating patients with cardiovascular disease. Electroacupuncture is a combination of traditional Chinese acupuncture and modern electrical techniques. The PC6 (Neiguan) acupoint is believed to influence cardiovascular function and treat a wide range of heart diseases, including angina pectoris, myocardial infarction, hypertension and hypotension.

According to traditional Chinese medicine theory, PC 6 (Neiguan) and LU 7 (Lieque) are important acupuncture points where two main meridians meet each other. LU 7 and LU 2 (Yunmen) belong to the same meridian. Three acupuncture points have coordinated effects and act together. These points are the most commonly used areas to treat heart diseases in China and other countries and have been selected as suitable points in studies.

DETAILED DESCRIPTION:
The study is a prospective, randomized and controlled study and will be conducted in patients who underwent cardiopulmonary bypass and coronary artery surgery.Randomized patients will be randomly divided into two groups as follows. Acupuncture group; Group A and Control group: Group C. In this study, the patients' age, gender, body mass index (BMI), smoking, comorbidities, left ventricular ejection/fraction (E/F), cardiopulmonary bypass time (CPBS, min), aortic cross-clamp time (ACCS, min). , operation duration, amount of cardioplegia, lowest body temperature will be recorded. Electroacupuncture will be applied to the patients for 30 minutes by the conductor of the study, who is an acupuncturist experienced in electroacupuncture, on the day before surgery and on the day of surgery.The placement of the needles will be applied to a depth of 1-2 cm, depending on the thickness of the local tissues, according to Traditional Chinese Medicine standards.The EA parameter will be set to a frequency of 2 HZ/100 HZ at a current that the patients' tolerance is best within the range of 0.5 mA to 1.2 mA and will be electrically stimulated for 30 minutes until the patient feels "Teh Chi" "heaviness, numbness and swelling". No acupuncture procedure will be applied to the patients in the control group.Routine anesthesia and surgery will be applied. All operations will be performed by the same surgical and anesthesia team. Patients will undergo radial artery catheterization and be monitored.Anesthesia will be provided using midazolam, fentanyl and rocuronium bromide. Sevoflurane will be used as an anesthetic agent for the maintenance of general anesthesia. Rocuronium bromide (0.6 mg.kg-1) will be administered every 30 minutes. A median sternotomy will be performed on each patient.Heparin will be administered at 300-500 units kg-1 and will be neutralized with 1-1.3 mg protamine sulfate. The type and amount of cardioplegia used will be recorded. During the procedure, an activated clotting time of >400 seconds and a mean arterial pressure (MAP) of >60 mmHg will be ensured. By applying PRAM, a minimally invasive advanced hemodynamic parameters monitoring system in our study (MostCare®, Vygon, Vytech), the data we will measure will be kept within reference ranges as much as possible. Noradrenaline, dopamine, dobutamine and glyceryl trinitrate (perlinganite) will be used to maintain within these reference ranges.Hemodynamic data we will measure by applying PRAM; Dicrotic Pressure, mean arterial pressure (MAP), stroke volume, cardiac output, systemic vascular resistance (SVR), cardiac cycle efficiency, the maximal slope of systolic upstroke (dp/dtmax), arterial elastance, pulse pressure variation, stroke volume variation, values. These values will be recorded as baseline values when the patients are taken to the operating table.In additionally, These values will be recorded at 10-20-30-40-50-60 minutes after the patient has undergone sternotomy and at 10-20-30-40-50-60 minutes after the patient leaves the pump.At these times, intra-group and inter-group comparisons will be made. During these time units, hemoglobin and hematocrit values will also be recorded.These values will be tried to be kept within the normal reference range. Intraoperative inotropic agent use scores will be calculated. In addition, preoperative heart rhythm (sinus or atrial fibrillation) and postoperative heart rhythm will be recorded.BIS score will be kept between 40-50. After the surgery, each patient will be taken to the cardiovascular surgery intensive care unit.

Blood samples for measurement of troponin I, ischemic modified albumin (IMA), interleukin 6, interleukin 10 will be taken from the radial artery before aortic cross-clamping (as baseline value before sternotomy) and at 1st hour, 6th hour, 12th hour, 24th hour and after removal of the aortic cross-clamp. The fluid, blood transfusion and platelet products taken throughout the operation will be recorded. The amount of blood planned to be taken in the study was determined to be at least 5 ml each time in order to study the relevant parameters. Considering that the patient will be hemodynamically supported during coronary bypass surgery, the total amount of blood to be taken during this time period related to the study is not expected to cause any undesirable changes in the patient's hemodynamic and biochemical aspects. Postoperative data; duration of mechanical ventilation in the intensive care unit (time intubated, min), duration of stay in the intensive care unit. Postoperative complications and the development of postoperative atrial fibrillation (AF) will be recorded. Inotropic agents used at 1 hour, 6th hour, 12th hour and 24th hour in the intensive care unit will be recorded and inotropic scores will be calculated.

According to the inotropic scoring method used in this study, it will be calculated as dopamine (x1), dobutamine (x1), amrinone (x1), epinephrine (x 100) and norepinephrine (x100). Again, total chest drainage volume and urine will be monitored in the intensive care unit, and the duration of intensive care stay (days) will be recorded. Blood samples will be frozen at -70°C until the plasma, separated after centrifugation, is assayed.

Troponin I concentrations will be measured quantitatively with a one-step enzyme immunoassay (Access AccuTnI assay system; Beckman-Coulter, Fullerton, CA) by individuals blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification III,
* 18-65 years old,
* Conscious Open,
* Participating in the study and giving permission to practice acupuncture,
* Does not require emergency or repeat surgery,
* Ejection/Fraction (E/F) ratio of 50-55%
* Patients extubated within 24 hours after transfer to intensive care

Exclusion Criteria:

* Patients who do not want to participate in the study,
* Patients with systemic diseases such as advanced liver, kidney and lung disease,
* Those with chronic inflammatory diseases (rheumatoid arthritis and psoriasis),
* Patients receiving immune systemic therapy,
* Patients with poor mental status,
* Patients with a history of epilepsy,
* Patients with pacemakers,
* Patients who have had heart surgery and emergency within the last month,
* Patients with atrial fibrillation,
* Patients who have atrial fibrillation and cannot be measured after coming off the pump,
* Patients who were not extubated within 24 hours after transfer to intensive care were excluded from the study.
* Additionally, patients receiving the antidiabetic sulfonylurea or glibenclamide were excluded because these agents have been shown to abolish the cardioprotective effect elicited by ischemic preconditioning.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Troponin I | At baseline levels, 1st hour, 6th hour, 12th hour, 24th hour changes after removal of the aortic cross-clamp,
  shows the myocardial injury

SECONDARY OUTCOMES:
Ischemic modified albumin (IMA) | At baseline levels, 1st hour, 6th hour, 12th hour, 24th hour changes after removal of the aortic cross-clamp,
  IMA occurs in hypoxic heart tissue through mechanisms related to muscle damage, decreased coronary blood flow, and modification of albumin by reactive oxygen species (ROS) increased by ischemic damage.
Interleukin 6 | At baseline levels, 1st hour, 6th hour, 12th hour, 24th hour changes after removal of the aortic cross-clamp,
  Interleukin 6 is an interleukin that acts as a pro-inflammatory cytokine
Interleukin 10 | At baseline levels, 1st hour, 6th hour, 12th hour, 24th hour changes after removal of the aortic cross-clamp,
  Interleukin 10 is an anti-inflammatory cytokine.
Dicrotic pressure | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  occurs during isovolumetric relaxation
mean arterial pressure | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  hemodynamic parameter
systemic vascular resistance | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  systemic vascular resistance is the resistance that must be overcome to push blood through the circulatory system and create blood flow
stroke volume | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  stroke volume is the volume of blood pumped from the left ventricle per beat
cardiac output | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  cardiac output is the volume of blood being pumped by a single ventricle of the heart
dp/dtmax | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  Change of left ventricular pressure over time
Cardiac cycle efficiency | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  Cardiac cycle efficiency provides a global assessment of total cardiovascular performance, measured in terms of energy expenditure.
Arterial elastance (Ea) | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  Arterial elastance is mainly related to the elasticity of the arterial system
Pulse pressure variation (PPV) | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  Dynamic fluid responsiveness parameter
Stroke Volume Variation (SVV) | Baseline changes after sternotomy at 10, 20, 30, 40, 50, 60 minutes and pump discontinuation at 10, 20, 30, 40, 50, 60 minutes
  Dynamic fluid responsiveness parameter

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Orak, Principal Investigator — Kahramanmaras Sutcu Imam University Faculty Medicine, anesthesiology and Reanimation Department
Locations (1):
- Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No